CLINICAL TRIAL: NCT02578745
Title: Prophylactic Negative Pressure Wound Therapy in Obese Women After Cesarean: a Pilot Randomized Trial
Brief Title: Prophylactic Incisional Care in Obese Women at Cesarean
Acronym: PICO-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB ID # 201508154
Record Dates: First submitted 2015-10-09; First posted 2015-10-19 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Wound Infections
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prophylactic NPWT (Experimental): Women assigned to prophylactic NPWT will have the PICO device applied and secured with fixation adhesion strips. The device will be monitored while the patient is in the hospital to confirm that it is functioning well. The device will be removed prior to discharge, typically on postoperative day 4.
  Interventions: Device: Prophylactic NPWT (PICO system)
- Standard Dressing (Active Comparator): Women assigned to standard care will receive routine postoperative wound dressing consisting of layers of gauze and adhesive tap. The dressing will be removed after 24 - 48 hours.
  Interventions: Other: Standard Dressing

INTERVENTIONS:
Device: Prophylactic NPWT (PICO system) — The PICO NPWT system is a small, lightweight (~126 grams), portable suction device consisting of an electric motor-driven vacuum pump connected to a proprietary super-absorbent adhesive dressing. It is supplied as a pump with two sterile dressing kits and two batteries. Different dressing sizes are available for transverse and vertical incisions ranging from 10 to 40 cm. The PICO pump maintains negative pressure of -80 mmHg (+/-20 mmHg) to the wound surface.
  Arms: Prophylactic NPWT
Other: Standard Dressing — Standard wound dressing consists of routine postoperative wound dressing consisting of layers of gauze and adhesive tape.
  Arms: Standard Dressing

SUMMARY:
Surgical site infections (SSIs) complicate 5 - 12% of cesareans. Negative pressure wound therapy (NPWT) - a closed, sealed system that applies negative pressure to the wound surface - has been used to treat open wounds since the late 1990s. Experimental evidence suggests NPWT promotes wound healing by removing exudate, approximating the wound edges, and reducing bacterial contamination. Although effectiveness of prophylactic NPWT is biologically plausible and non-randomized studies suggest benefit in reducing SSIs, good quality data is lacking. The objective of this pilot randomized controlled trial of 120 patients to test the hypothesis that prophylactic NPWT will reduce SSIs and other wound complications after cesarean in obese women. The investigators will randomly assign obese women undergoing cesarean delivery to Standard dressing or prophylactic NPWT with the PICO system after skin closure. The primary outcome will be a composite of superficial or deep SSIs per Centers for Disease Control and Prevention (CDC) criteria and other wound complications (separation, hematoma, seroma) after cesarean.

Secondary outcomes will include wound dehiscence (≥2 cm); hematoma; seroma; composite of wound complications; patient pain and satisfaction scores; physician office visit or emergency department (ED) visits for SSIs; and hospital readmission for wound complications.

DETAILED DESCRIPTION:
Overview of the Proposed Trial

This will be a pilot randomized controlled trial. The investigators chose a randomized controlled trial, the 'gold standard' of clinical research design, with the goal of obtaining the highest quality evidence to inform clinical practice. Randomly allocating subjects to different interventions minimizes selection bias and results in groups that are comparable with regards to important confounding variables, both measured and unmeasured. Additionally, the broad inclusion criteria, simplicity of the interventions, and evaluation of effects of typical use of prophylactic NPWT make this a pragmatic trial. The investigators will follow the Consolidated Standards of Reporting Trials (CONSORT) guidelines in the conduct and reporting of this trial. We will use computer-generated block randomization stratified by study site and BMI category to assign participants to the two interventions. All subjects will receive standard infection prevention measures including skin antisepsis and weight-adjusted prophylactic antibiotics. Analysis will follow the intention-to-treat principle. The use of broad inclusion criteria and intention-to-treat analysis will allow a more conservative estimate of the effect of prophylactic NPWT and allow a better estimate of effectiveness and public health implications of practice change than would pure estimate of efficacy alone.

Conduct of the Trial Recruitment of study subjects: All women admitted to the labor and delivery units of the participating medical centers will be screened against inclusion and exclusion criteria. Eligible subjects will be approached by trained research staff for written consent to participate in the study. Subjects will be randomized only when the decision is made for cesarean delivery.

Randomization and allocation concealment: Enrolled subjects will be randomly assigned in a 1:1 ratio to NPWT or standard care using a computer-generated random sequence generated by the study statistician. A subject's group assignment will be revealed only after the decision is made to perform cesarean delivery.

Blinding: Although blinding of both subjects and physicians would be ideal, blinding is not possible in this trial. We will minimize systematic bias by applying the same standard infection prevention measures in all patients at each site. Further, the research personnel collecting outcomes data will be blinded to the group assignments of the subjects after the standard dressing or NPWT device have been removed. Importantly, diagnosis of the primary outcome will be objectively reviewed centrally by the PI in a blinded fashion using to CDC criteria.

Interventions: The interventions to be compared in this trial are standard care versus prophylactic NPWT after skin closure:

1. Standard care: Women assigned to standard care will receive routine postoperative wound dressing consisting of layers of gauze and adhesive tap. The dressing will be removed after 24 - 48 hours.
2. Prophylactic NPWT: Women assigned to prophylactic NPWT will have the PICO device applied and secured with fixation adhesion strips. The device will be monitored while the patient is in the hospital to confirm that it is functioning well. The device will be removed prior to discharge, typically on postoperative day 4.

Rationale for choosing PICO: There are no head-to-head trials of the two FDA-cleared prophylactic NPWT devices, and the preliminary data do not suggest one is superior to the other. However, there is a large price difference: $200 per PICO unit and $500 per Prevena unit. The investigators chose the less expensive device.

Data Collection: The investigators will collect detailed antepartum, intrapartum, and postpartum information from study participants. Relevant data will be collected initially to assess eligibility. Complete baseline information and outcome data will be collected by trained study nurses by direct interview and chart review.

Hypothesis Testing Primary Aim: Determine the effectiveness of prophylactic NPWT in reducing the rate of SSIs and other wound complications after cesarean in obese women.

Hypothesis: Obese women will have lower rates of SSIs and other wound complications after cesarean with use of prophylactic NPWT than with standard care.

Primary outcome: The primary outcome for the trial is superficial or deep SSIs and other wound complications (separation, hematoma, seroma) after cesarean. This will be defined according to CDC criteria as infections at the surgical site occurring within 30 days of cesarean delivery, and classified as superficial, deep, or organ/space occupying. We will use active surveillance for SSIs including one patient phone call by the research coordinator within 30 days after surgery. The PI will blindly review de-identified inpatient and outpatient records of all subjects with suspected SSIs against CDC criteria to ensure standard diagnosis and classification.

Secondary outcomes: Wound dehiscence (≥2 cm); hematoma; seroma; composite of wound complications; patient pain and satisfaction scores (on a scale of 0 to 10) at discharge and postoperative day 14 (±2 days) and 28 (±2 days); physician office visit or ED visits for SSIs; and hospital readmission for SSIs.

Sample size calculation: The sample size for this pilot trial is 120; 60 in the prophylactic NPWT group and 60 in the standard treatment group. We estimated the sample size for the trial assuming a baseline SSI and wound complication rate of 24% based on a recent trial at our institution, and we a clinically significant 75% reduction effect size based on a recently published study.

CDC Criteria for defining and classifying surgical site infections (SSIs):

1. Superficial incisional (wound) infection infection occurs within 30 days after operative procedure; AND involves only skin and subcutaneous tissue of the incision; AND patient has at least one of the following:

   1. purulent drainage from the superficial incision,
   2. organisms isolated from an aseptically-obtained culture from the superficial incision or subcutaneous tissue,
   3. superficial incision that is deliberately opened by a surgeon, attending physician or other designee and is culture-positive or not cultured; and patient has at least one of the following signs or symptoms: pain or tenderness; localized swelling; erythema; or heat. A culture-negative finding does not meet this criterion,
   4. diagnosis of a superficial incisional SSI by the surgeon or attending physician or other designee.
2. Deep incisional (wound) infection

   Infection occurs within 30 days of operative procedure; AND involves deep soft tissues of the incision (e.g., fascial and muscle layers); AND patient has at least one of the following:
   1. purulent drainage from the deep incision,
   2. a deep incision that spontaneously dehisces, or is deliberately opened or aspirated by a surgeon, attending physician or other designee and is culture-positive or not cultured; and patient has at least one of the following signs or symptoms: fever (>38°C), localized pain, or tenderness. A culture-negative finding does not meet this criterion,
   3. an abscess or other evidence of infection involving the deep incision that is detected on gross anatomical or histopathologic exam, or imaging test.
3. Organ/Space (endometritis, abscess)

Infection occurs within 30 days of operative procedure; AND infection involves any part of the body deeper than the fascial/muscle layers, that is opened or manipulated during the operative procedure; AND patient has at least one of the following:

1. purulent drainage from a drain that is placed into the organ/space (e.g., closed suction drainage system, open drain, T-tube drain, CT-guided drainage),
2. organisms isolated from an aseptically-obtained culture of fluid or tissue in the organ/space,
3. an abscess or other evidence of infection involving the organ/space that is detected on gross anatomical or histopathologic exam, or imaging test; AND meets at least one criterion for a specific organ/space infection site.

Secondary Aim 1: Assess the safety of prophylactic NPWT in obese women as measured by frequency of adverse events including skin blisters, erythema, wound bleeding and prolonged wound drainage.

Hypothesis: The rate of adverse events will not be significantly higher with use of prophylactic NPWT than with standard care.

Outcomes for secondary aim 1: Composite of adverse events potentially attributable to NPWT including skin blisters, erythema, wound bleeding, and prolonged (>7 days) wound drainage.

Rationale: NPWT has been associated with adverse events including skin blisters, wound bleeding, and prolonged wound drainage. A high rate of skin blisters was reported when NPWT was used after orthopedic surgery. This was attributed to use of the adhesive dressing in the setting of marked swelling and edema. Although the adverse events noted with NPWT after cesarean have generally been minor and were comparable in frequency to use of standard dressing, it is essential to characterize the frequency of these events to permit risk-benefit counseling of patients.

Secondary Aim 2: Determine the effect of prophylactic NPWT on the frequency and identity of bacteria, including antibiotic-resistant organisms, isolated from SSIs after cesarean in obese women.

Hypothesis: Prophylactic NPWT will be associated with a reduction in the rate of positive wound cultures and antibiotic-resistant bacteria isolated from SSIs after cesarean.

Outcomes for secondary aim 2: Rate of positive wound cultures and proportion of specific organisms, especially drug-resistant bacteria (e.g. MRSA) isolated from SSIs after cesarean.

Wound cultures and antimicrobial sensitivity testing: Physicians will follow clinical protocols that warrant collection of swabs from all accessible SSIs for routine aerobic and anaerobic cultures.

Data Analysis Plan Overview: Data analyses will adhere closely to the CONSORT guidelines. Analyses will follow the intention-to-treat principle in which subjects will be analyzed in the group to which they were randomized, regardless of whether or not they received the assigned intervention.

Primary Analysis: Descriptive statistics will characterize the group of individuals recruited and investigate comparability of the two groups at baseline. Formal statistical testing will be limited to selected baseline characteristics considered to be prognostic factors for the primary outcome such as emergent cesarean, type of skin incision, and prolonged rupture of membranes. The categorical prognostic factors will be compared between trial groups by using the Fisher's exact test. Continuous prognostic factors will be compared using the Mann-Whitney U test.

The primary outcome and other categorical secondary outcomes will be compared between intervention groups by using the Cochran-Mantel-Haenszel test.The investigators will calculate common relative risks and 95% confidence intervals associated with the primary and secondary outcomes. The investigators will also conduct time-to-event analyses by using Kaplan Meier and Cox regression models to examine the pattern of SSIs in the two groups.

Secondary Analyses: The investigators will perform other analyses aimed at obtaining adjusted estimates of treatment effectiveness, adjusting for baseline subject characteristics (covariates). The objectives of these analyses are to estimate the influence of covariates on the outcome and to use covariates to improve the estimated difference between treatment groups. Stepwise logistic regression models will be used to identify and estimate the effect of multiple prognostic factors on the probability of SSI and other categorical outcomes. Interaction tests will be used to determine whether the effectiveness of prophylactic NPWT differs across these subgroups such as BMI category and type of skin incision. These secondary analyses will be considered exploratory.

Safety monitoring

The interventions compared in this trial are both currently used in clinical obstetric practice. Further, the adverse events reported with use of prophylactic NPWT at cesarean were minor and their frequency was comparable to rates with standard dressing. Therefore, no serious or life-threatening adverse events are expected. Nonetheless, the following measures will be taken to monitor and investigate adverse events:

1. Adverse events reporting: Detailed information concerning adverse events will be collected and evaluated throughout the trial. If a participant develops an adverse event, the participant's physician and PI will ascertain the safety of continuing the intervention.
2. Interim analyses: The investigators anticipate one interim analyses after 60 patients have recruited. Although early stopping decisions cannot be based purely on a mathematical stopping rule, we will use the Haybittle-Peto stopping rule as a guide. Under this rule, the interim analyses of the primary outcome would have to demonstrate an extreme difference between groups (P <0.001) to justify premature disclosure. This rule has the advantages that the exact number of interim analyses need not be specified in advance and the overall type I error is preserved at 0.05; therefore, samples size adjustment is not needed.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≥23weeks
* BMI≥30 at the time of delivery
* Planned or unplanned cesarean delivery (procedure in which NPWT is being tested)

Exclusion Criteria:

* Non-availability for postoperative follow-up (follow-up is needed to ascertain study outcomes)
* Contraindication to NPWT applicable to women undergoing cesarean (device will not be used in patients with contraindications): Pre-existing infection around incision site, Bleeding disorder, Therapeutic anticoagulation, Allergy to any component of the dressing (e.g. silicone, adhesive tape)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Methodius G Tuuli, MD, MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bullough L, Spruce P. Removing all barriers: a 10-patient evaluation in the acute care setting. Br J Nurs. 2013 Nov 14-27;22(20):S38, S40-4. doi: 10.12968/bjon.2013.22.Sup20.S38. PMID 24225510
- [Background] Mark KS, Alger L, Terplan M. Incisional negative pressure therapy to prevent wound complications following cesarean section in morbidly obese women: a pilot study. Surg Innov. 2014 Aug;21(4):345-9. doi: 10.1177/1553350613503736. Epub 2013 Sep 20. PMID 24056202
- [Background] Darouiche RO, Wall MJ Jr, Itani KM, Otterson MF, Webb AL, Carrick MM, Miller HJ, Awad SS, Crosby CT, Mosier MC, Alsharif A, Berger DH. Chlorhexidine-Alcohol versus Povidone-Iodine for Surgical-Site Antisepsis. N Engl J Med. 2010 Jan 7;362(1):18-26. doi: 10.1056/NEJMoa0810988. PMID 20054046
- [Background] Swift SH, Zimmerman MB, Hardy-Fairbanks AJ. Effect of Single-Use Negative Pressure Wound Therapy on Postcesarean Infections and Wound Complications for High-Risk Patients. J Reprod Med. 2015 May-Jun;60(5-6):211-8. PMID 26126306
- [Background] Bullough, L, Wilkinson, D., Burns, S, Wan, L, Changing wound care protocols to reduce postoperative caesarean section infection and readmission, Wounds , 2014 (10), 1 : 72 - 76. 46

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 120 patients from October 2015 to April 2016 at Washington University Medical Center
Pre-assignment Details: We enrolled patients undergoing scheduled or emergency cesarean delivery.
Groups:
- Prophylactic NPWT: Women assigned to prophylactic NPWT had the PICO device applied and secured with fixation adhesion strips. The device was monitored while the patient was in the hospital to confirm that it wass functioning well. The device will be removed prior to discharge, typically on postoperative day 4.
  Prophylactic NPWT (PICO system): The PICO NPWT system is a small, lightweight (~126 grams), portable suction device consisting of an electric motor-driven vacuum pump connected to a proprietary super-absorbent adhesive dressing. It is supplied as a pump with two sterile dressing kits and two batteries. Different dressing sizes are available for transverse and vertical incisions ranging from 10 to 40 cm. The PICO pump maintains negative pressure of -80 mmHg (+/-20 mmHg) to the wound surface.
- Standard Dressing: Women assigned to standard care had routine postoperative wound dressing consisting of layers of gauze and adhesive tap. The dressing was removed after 24 - 48 hours.
  Standard Dressing: Standard wound dressing consists of routine postoperative wound dressing consisting of layers of gauze and adhesive tape.
Period: Overall Study
Arm/Group | Prophylactic NPWT | Standard Dressing
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Prophylactic NPWT: Women assigned to prophylactic NPWT had the PICO device applied and secured with fixation adhesion strips. The device was monitored while the patient is in the hospital to confirm that it is functioning well. The device was removed prior to discharge, typically on postoperative day 4.
  Prophylactic NPWT (PICO system): The PICO NPWT system is a small, lightweight (~126 grams), portable suction device consisting of an electric motor-driven vacuum pump connected to a proprietary super-absorbent adhesive dressing. It is supplied as a pump with two sterile dressing kits and two batteries. Different dressing sizes are available for transverse and vertical incisions ranging from 10 to 40 cm. The PICO pump maintains negative pressure of -80 mmHg (+/-20 mmHg) to the wound surface.
- Total: Total of all reporting groups
Arm/Group | Prophylactic NPWT | Standard Dressing | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (6.6) | 28.7 (5.0) | 29.0 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 60 | 120
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 57 | 58 | 115
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 40 | 36 | 76
  White | 20 | 23 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 39.2 (9.2) | 40.7 (8.6) | 39.9 (8.9)
Scheduled cesarean [Count of Participants; unit: Participants] | 56 | 56 | 112

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite Surgical Site Infection (SSI) or Other Wound Complication.
Description: Superficial or deep SSIs or other wound complications (separation, hematoma, seroma) after cesarean. SSI will be defined according to the Centers for Disease Control (CDC) criteria as infections at the surgical site occurring within 30 days of cesarean delivery, and classified as superficial, deep, or organ/space occupying.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Prophylactic Negative Pressure Wound Therapy (NPWT): Women assigned to prophylactic NPWT had the PICO device applied and secured with fixation adhesion strips. The device was monitored while the patient is in the hospital to confirm that it is functioning well. The device was removed prior to discharge, typically on postoperative day 4.
  Prophylactic NPWT (PICO system): The PICO NPWT system is a small, lightweight (~126 grams), portable suction device consisting of an electric motor-driven vacuum pump connected to a proprietary super-absorbent adhesive dressing. It is supplied as a pump with two sterile dressing kits and two batteries. Different dressing sizes are available for transverse and vertical incisions ranging from 10 to 40 cm. The PICO pump maintains negative pressure of -80 mmHg (+/-20 mmHg) to the wound surface.
Arm/Group | Prophylactic Negative Pressure Wound Therapy (NPWT) | Standard Dressing
Number analyzed (Participants) | 60 | 60
Participants | 5 | 3
Statistical Analysis 1: Comparison: Prophylactic Negative Pressure Wound Therapy (NPWT) vs Standard Dressing; Test type: Superiority; p = 0.72, Chi-squared; Risk Ratio (RR) = 1.67, 95% CI 2-sided [.42 to 6.67]

2. Secondary Outcome: Number of Participants With Any COMPONENT of SSI or Composite Wound Complication
Description: Proportion of Participants with Surgical site infection; Proportion of Participants with wound separation; Proportion of participants with hematoma; Proportion of participants with seroma.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic NPWT | Standard Dressing
Number analyzed (Participants) | 60 | 60
Participants | 5 | 3
Statistical Analysis 1: Comparison: Prophylactic NPWT; Test type: Superiority; p = 0.72, Chi-squared; Risk Ratio (RR) = 1.67, 95% CI 2-sided [.42 to 6.67]

3. Secondary Outcome: Pain Score on a 0 to 10 on Likert Scale
Description: Participant pain scores on postoperative day 2 on a 0 (minimum) to 10 (maximum) 0n Likert Scale, where 0 is no pain and 10 is the worse pain. Higher score means worse outcome
Time Frame: Postoperative days 2
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Prophylactic NPWT | Standard Dressing
Number analyzed (Participants) | 60 | 60
units on a scale | 0 [0 to 1] | 1 [1 to 3]
Statistical Analysis 1: Comparison: Prophylactic NPWT vs Standard Dressing; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Participants With Positive Wound Culture
Description: Rate of positive wound culture in participants with SSI after cesarean.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic NPWT | Standard Dressing
Number analyzed (Participants) | 60 | 60
Participants | 0 | 0
Statistical Analysis 1: Comparison: Prophylactic NPWT vs Standard Dressing; Test type: Superiority; p > 0.99, Chi-squared

5. Secondary Outcome: Number of Participants With Methicillin-resistant Staphylococcus Aureus.
Description: Rate of methicillin-resistant Staphylococcus aureus in patients with SSI after cesarean.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic NPWT | Standard Dressing
Number analyzed (Participants) | 60 | 60
Participants | 0 | 0
Statistical Analysis 1: Comparison: Prophylactic NPWT vs Standard Dressing; Test type: Superiority; p > 0.99, Chi-squared

6. Secondary Outcome: Number of Participants With Any Prophylactic Negative Pressure-related Adverse Events.
Description: Rate of composite of adverse events potentially attributable to NPWT including skin blisters, erythema, wound bleeding.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic NPWT | Standard Dressing
Number analyzed (Participants) | 60 | 60
Participants | 2 | 0
Statistical Analysis 1: Comparison: Prophylactic NPWT vs Standard Dressing; Test type: Superiority; p = 0.50, Chi-squared

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Prophylactic NPWT | Standard Dressing
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 2/60 | 0/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylactic NPWT (N=60) | Standard Dressing (N=60)
Pruiritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes